CLINICAL TRIAL: NCT06878482
Title: Effect of Increasing Blood Flow by Botulinum Toxin Local Injection for Severe Peripheral Artery Occlusive Disease: Preliminary Report
Brief Title: Effect of Blood Flow by Botulinum Toxin Injection for Severe Peripheral Artery Occlusive Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hii Sun Jeong, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9-2023-0006
Record Dates: First submitted 2024-01-22; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Ulcer of Lower Extremity; Wound; Botulinum Toxins, Type A; Blood Circulation
Keywords: Botulinum Toxins, Type A; Wound; Chronic Ulcer of Lower Extremity; Blood Circulation
MeSH Terms: conditions — Wounds and Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Botulinum toxin A (Experimental): Single group(Botulinum toxin A) Open label
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — subcutaneous injection of Botulinum toxin A

SUMMARY:
The purpose of this study is to investigate the effect of subcutaneous injection of botulinum toxin A on wound healing caused by lower extremity ischemia.

DETAILED DESCRIPTION:
Tissues below the calf are governed by blood flow from the anterior tibial artery, peroneal artery, and posterior tibial artery. When an ulcer occurs due to acute lower extremity ischemia, one of the three blood vessels is blocked by a blood clot, or when the blood vessel is narrowed due to perivascular inflammation, such as Buerger's disease, it occurs in a subacute or chronic form. In particular, in the case of elderly patients with ulcers or diabetic feet due to lower extremity ischemia, the symptoms are often worsened by chronic narrowing of blood vessels due to arteriosclerosis or blockage by blood clots. To treat this, prostaglandin or antithrombotic drugs are taken, and blood flow is resumed through stent surgery, but in the lower extremities, the recurrence rate is relatively high because the blood vessels are smaller than the iliac artery, femoral artery, and popliteal artery.

Botulinum toxin is known to have a positive effect on wound healing and blood flow improvement. Botulinum toxin has been published several times in papers showing its spasmolytic effect by participating in the radiographic hip osteoarthritis Ras homolog A (RhoA)/Rock-assisted protein kinase (ROCK) pathway. In addition, botulinum toxin has a vasodilating effect related to the calcitonin gene-related peptide (CGRP) pathway, and is involved in increasing vascular endothelial growth factor (VEGF) from NO-mediated angiogenesis, inhibiting vasoconstriction, increasing blood flow rate, and promoting angiogenesis.

In this study, in patients with chronic wounds on the feet, whose lower extremity blood vessels circulate mainly through collateral circulation, subcutaneous injection of Botulinum toxin in and around the wound improves blood flow around the wound and confirms the degree of wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years old
2. Patients who have a lower extremity wound among those who have been diagnosed with moderate or severe lower extremity ischemia
3. Patients who are unable to perform additional procedures (angioplasty, etc.) by performing peripheral vascular examination and CT angiography
4. Wound size ≥ 1x1cm2 to ≤ 3x3cm2
5. Patients who can follow the clinical trial procedure well and abide by the visit schedule
6. Written informed consent to participate in the study after having fully understood the contents of the protocol and restrictions.

Exclusion Criteria:

1. Patients with diseases that can affect neuromuscular function, such as myasthenia gravis, Eaton-Lamberton syndrome, amyotrophic lateral sclerosis, and motor neuropathy
2. Within 4 weeks before screening, aminoglycoside antibiotics, curare-like agents, or drugs that inhibit neuromuscular function (muscle relaxants, anticholinergics, benzodiazepines, benzamides, tetracyclines, Rinco Those who have taken mycin antibiotics, etc.)
3. Those taking aspirin, NSAIDs or anticoagulants within 7 days before screening
4. Those who have received botulinum toxin preparations within 3 months before screening
5. Angiography or CT angiography If one or more of the three major blood vessels in the lower extremity are open
6. Cases in which blood flow to the lower extremities can be preserved by performing balloon angioplasty even if all three major blood vessels in the lower extremity are blocked
7. Those who are currently taking steroids or immunosuppressants that affect wounds, or those who have taken them within one month of screening
8. Those who have applied injection drugs or wound coverings that help improve wounds within 1 week of screening
9. Women who are pregnant, lactating, planning to become pregnant during the clinical period, or women of childbearing age who are not using available contraceptive methods (women of childbearing age must be negative in the pregnancy test prior to injection).
10. Those who are allergic or sensitive to botulinum toxin
11. Those who have participated in another clinical trial within 30 days before screening or those who have not passed the half-life of the investigational product of the clinical trial that they participated in, whichever is longer.
12. Those who are not suitable for this clinical trial under the judgment of other investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in tcPO2(mmHg) measurement within the edge of 1cm Diabetic foot wound at 7 days and 14 days after IP compared to baseline(Pre-administration IP) | Baseline/7days after IP/14days after IP
  tcPO2 measurement

SECONDARY OUTCOMES:
Change in color-graded amount(using Thermal Imaging Camera) within Diabetic foot wound at 7 days and 14 days after IP compared to baseline(Pre-administration IP) | Baseline/7days after IP/14days after IP
  color-graded amount(using Thermal Imaging Camera)
Changes in wound quality and area in photographs at 7 days and 14 days after IP compared to baseline(Pre-administration IP) | Baseline/7days after IP/14days after IP
  wound quality and area in photographs(Digital Camera)

CONTACTS AND LOCATIONS:
Overall Officials: Hiisun J, Dr, Principal Investigator — Yonsei University College of Medicine, Yongin Severance
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Roh TS, Jung BK, Yun I, Lew DH, Kim YS. Effect of botulinum toxin A on vasoconstriction and sympathetic neurotransmitters in a murine random pattern skin flap model. Wound Repair Regen. 2017 Jan;25(1):75-85. doi: 10.1111/wrr.12501. Epub 2017 Jan 5. PMID 27997734

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT06878482/Prot_SAP_000.pdf